CLINICAL TRIAL: NCT03859024
Title: Efficacy of Opioid-limiting Pain Management Protocol in Men Undergoing Urethroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Adam Baumgarten, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002992
Record Dates: First submitted 2019-02-27; First posted 2019-03-01 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Urethral Stricture
Keywords: anterior urethroplasty; pain management; postoperative pain; opioid use
MeSH Terms: conditions — Pain, Postoperative; Urethral Stricture; Agnosia | interventions — Oxycodone; Acetaminophen; Gabapentin; Celecoxib; Bupivacaine; Ibuprofen; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard Protocol (Active Comparator): Patients will receive the historical standard for pain management, which may include narcotics during and after surgery. Postoperative prescriptions ibuprofen 800 mg, and acetaminophen 1000 mg to be taken on a scheduled basis then as needed. Another prescription for oxycodone will be given to be used only if needed.
  Interventions: Drug: Oxycodone; Drug: Acetaminophen; Drug: Ibuprofen 800 mg
- Enhanced Recovery Protocol (Experimental): A combination regimen of acetaminophen, Celebrex and gabapentin pre-op, with 30 mL of 0.5% bupivacaine and 4 mg of dexamethasone given as a perineal nerve block at the time of urethroplasty surgery. Narcotics will be administered judiciously and ass seen fit by the anesthesia and/or surgical teams. Postoperative prescriptions ibuprofen 800 mg, and acetaminophen 1000 mg to be taken on a scheduled basis then as needed. Another prescription for oxycodone will be given to be used only if needed.
  Interventions: Drug: Oxycodone; Drug: Acetaminophen; Drug: Gabapentin; Drug: celebrex; Drug: Bupivacaine; Drug: Ibuprofen 800 mg; Drug: Dexamethasone

INTERVENTIONS:
Drug: Oxycodone — oxycodone tablet
  Other Names: oxycontin
Drug: Acetaminophen — acetaminophen tablet
  Other Names: tylenol
Drug: Gabapentin — gabapentin tablet
  Other Names: neurontin
  Arms: Enhanced Recovery Protocol
Drug: celebrex — Celebrex tablet
  Other Names: celecoxib
  Arms: Enhanced Recovery Protocol
Drug: Bupivacaine — bupivacaine injection
  Other Names: marcaine, exparel
  Arms: Enhanced Recovery Protocol
Drug: Ibuprofen 800 mg — ibuprofen tablet
  Other Names: advil, motrin
Drug: Dexamethasone — Dexamethasone injection
  Other Names: decadron, ozurdex
  Arms: Enhanced Recovery Protocol

SUMMARY:
The investigator's study aims to see if an enhanced recovery regimen of pain medications before and during surgery will decrease the use and risk of opioid pain medications as well as improve pain control in anterior urethroplasty patients. Participants will be randomized to one of two pain regimens (enhanced recovery regimen vs standard regimen).

DETAILED DESCRIPTION:
The purpose of this study is to assess the difference in narcotics usage between two different pain management protocols after urethroplasty. Management at the current time varies between giving intraoperative painkillers along with peripheral nerve blocks in some patients, while others do not receive this protocol. In this study, one group will continue the historical standard of care of the hospital, receiving postoperative nonsteroidal anti-inflammatory drugs (NSAIDs) and narcotics for pain control. The other group will utilize a protocol to lower narcotics usage, including acetaminophen, gabapentin, Celebrex, and local anesthetic (bupivacaine) in an attempt to reduce the usage of narcotics postoperatively. Given the heightened concern over narcotic usage by postoperative patients, including the risk of chronic usage by even young patients, the objective will be to assess if using this protocol as a new standard can limit the need for postoperative narcotics prescriptions.

In related urological procedures, bupivacaine injections given before surgeries have been shown to significantly lower pain scores after surgery for patients undergoing penile prosthesis. The University of Alabama at Birmingham has also been using an Enhanced Recovery After Surgery (ERAS) protocol, a multimodal presurgical care pathway designed to achieve early recovery after surgical procedures, for cystectomy and seen reduced narcotic usage among those patients.

This study would potentially help determine a new pain management protocol for urology patients undergoing anterior urethroplasty that is both more effective and less risky.

ELIGIBILITY:
Inclusion Criteria:

* Men greater than 18 years of age who are scheduled for anterior urethroplasty surgery

Exclusion Criteria:

* Any patient not classified as a II or III on the American Society of Anesthesiologists (ASA) physical status classification system.
* General anesthesia or neuraxial anesthesia with epidural used as anesthetic techniques
* Allergy/intolerance to local anesthetic or steroids
* Pre-existing neurological and/or anatomical deficit that would preclude regional block
* Coexisting coagulopathy such as hemophilia or von Willebrand Disease
* BMI greater than 40 or less then 20
* History of intravenous drug or opioid abuse
* History of opioid use within a week prior to urethroplasty
* History of any chronic pain syndrome
* Posterior urethroplasty
* Patients with chronic kidney disease
* Patients allergic to NSAIDs
* Patients requiring more than one buccal graft harvest
* Patients with graft urethroplasty with site other than buccal
* Patients with a history of previous urethroplasty

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Selph, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama of Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Protocol | Enhanced Recovery Protocol
Started | 23 | 25
Completed | 23 | 24
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Protocol | Enhanced Recovery Protocol | Total
Number analyzed (Participants) | 23 | 25 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 21 | 41
  >=65 years | 3 | 4 | 7
Age, Continuous [Mean (Full Range); unit: years] | 50 [28 to 80] | 50 [21 to 80] | 50 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 23 | 25 | 48
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Participant Pain Control: Numerical Rating Scale (NRS)
Description: Self-report via pain score on the Numerical Rating Scale (NRS) for pain, an 11-point scale for patient self-reporting of pain. A rating of 0 equates to no pain, 1-3 equates to mild pain, 4-6 equates to moderate pain, and 7-10 equates to severe pain. Assessment will occur at clinic visit, at pre-op visit, in pre-op holding before surgery, per anesthesia protocol after surgery in recovery and discharge unit, and at postoperative visit
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Standard Protocol | Enhanced Recovery Protocol
Number analyzed (Participants) | 23 | 24
score on a scale | 1.2 [0 to 10] | .625 [0 to 10]

2. Primary Outcome: Opioid Medication Use
Description: Amount of opioid medication used, based on return pill count at postoperative visit.
Time Frame: 3 weeks
Measure: Mean (Full Range); unit: pill count
Arm/Group | Standard Protocol | Enhanced Recovery Protocol
Number analyzed (Participants) | 23 | 24
pill count | 5.14 [0 to 14] | 4.96 [0 to 14]

ADVERSE EVENTS:
Time Frame: 3 weeks
Arm/Group | Standard Protocol | Enhanced Recovery Protocol
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/25
Other Adverse Events (participants affected / at risk) | 0/23 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-10-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03859024/Prot_000.pdf